CLINICAL TRIAL: NCT03264066
Title: A Phase II, Open-Label, Multicenter, Multicohort Study to Investigate the Efficacy and Safety of Cobimetinib Plus Atezolizumab in Patients With Solid Tumors
Brief Title: A Study to Investigate the Efficacy and Safety of Cobimetinib Plus Atezolizumab in Participants With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO39760; 2017-000794-37 (EudraCT Number)
Record Dates: First submitted 2017-08-17; First posted 2017-08-28 (Actual); Results first posted 2021-03-01 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumors
MeSH Terms: interventions — cobimetinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 - SCCHN - Treatment Naive (Experimental): In participants with recurrent or advanced / metastatic SSCHN who are anti-PD-1 and anti-PD-L1 treatment naive, cobimetinib will be administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Cohort 2 - UC - Treatment Naive (Experimental): In participants with advanced / metastatic UC who are anti-PD-1 and anti-PD-L1 treatment naive, cobimetinib will be administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Cohort 3 - RCC - Treatment Naive (Experimental): In participants with metastatic RCC who are anti-PD-1 and anti-PD-L1 treatment naive, cobimetinib will be administered at the approved dose and schedule of 60 milligrams (mg) once daily (QD) for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Cohort 4 - SCCHN - Previous Treatment Exposure (Experimental): In participants with SCCHN whose disease has progressed while receiving anti-PD-1 or anti-PD-L1 therapy, cobimetinib will be administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Cohort 5 - UC - Previous Treatment Exposure (Experimental): In participants with UC whose disease has progressed while receiving anti-PD-1 or anti-PD-L1 therapy, cobimetinib will be administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Cohort 6 - RCC - Previous Treatment Exposure (Experimental): In participants with RCC whose disease has progressed while receiving anti-PD-1 or anti-PD-L1 therapy, cobimetinib will be administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Cohort 7 - Biopsy Cohort (Experimental): In participants with solid non-melanoma, non- hematologic tumors who previously developed primary or secondary resistance to an anti-PD-1 or anti-PD-L1 agent, cobimetinib will be administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle. The first dose of atezolizumab of 840 mg by IV infusions on Day 15 of Cycle 1. Thereafter, they will receive atezolizumab 840 mg IV infusion Q2W on Days 1 and 15 of Cycle 2 and all subsequent cycles.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab Cohort 7

INTERVENTIONS:
Drug: Cobimetinib — Participants will receive cobimetinib 60 mg (3 tablets of 20 mg each) orally once a day on Days 1-21 of each 28-day cycle.
  Other Names: Cotellic
Drug: Atezolizumab — Atezolizumab will be given at a fixed dose of 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
  Other Names: Tecentriq
  Arms: Cohort 1 - SCCHN - Treatment Naive; Cohort 2 - UC - Treatment Naive; Cohort 3 - RCC - Treatment Naive; Cohort 4 - SCCHN - Previous Treatment Exposure; Cohort 5 - UC - Previous Treatment Exposure; Cohort 6 - RCC - Previous Treatment Exposure
Drug: Atezolizumab Cohort 7 — Only for participants in cohort 7, the first dose of atezolizumab of 840 mg will be given by IV infusion on Day 15 of Cycle 1; thereafter, they will receive atezolizumab 840 mg IV infusion Q2W on Days 1 and 15 of Cycle 2 and all subsequent cycles.
  Other Names: Tecentriq
  Arms: Cohort 7 - Biopsy Cohort

SUMMARY:
This is a study to evaluate the efficacy, safety, and pharmacokinetics of cobimetinib plus atezolizumab in participants with advanced solid tumors including the following cohorts: squamous cell carcinoma of the head and neck (SCCHN), urothelial carcinoma (UC), and renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Age ≥18 years
* Ability to comply with the study protocol, in the investigator's judgment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Life expectancy ≥3 months, as determined by the investigator
* Adequate hematologic and end-organ function

Cancer-Related Inclusion Criteria:

* Patients must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) scan per RECIST v1.1.
* Availability to provide a representative tumor specimen biopsy
* Evidence of tumor progression on or after the last treatment regimen received and within 6 months prior to study enrollment
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a non-hormonal contraceptive method with a failure rate of <1% per year during the treatment period and for at least 5 months after the last dose of atezolizumab and within 3 months after the last dose of cobimetinib
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm during the treatment period and for at least 3 months after the last dose of cobimetinib

Exclusion Criteria:

General Exclusion Criteria:

* Inability to swallow medications
* Malabsorption condition that would alter the absorption of orally administered medications
* Poor peripheral venous access
* Prior treatment with cobimetinib or a MEK inhibitor
* Prior treatment with T-cell co-stimulating or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with investigational therapy within 14 days prior to initiation of study treatment
* Any anti-cancer therapy, including chemotherapy or hormonal therapy, within 2 weeks prior to initiation of study treatment
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceutical agents produced in Chinese hamster ovary cells or any component of the atezolizumab formulation, or any component of the cobimetinib formulation
* History of serous retinopathy, retinal vein occlusion (RVO), or evidence of ongoing serous retinopathy or RVO at baseline
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage more than once every 28 days
* Uncontrolled hypercalcemia (ionized calcium >1.5 millimoles per liter [mmol/L], calcium >12 milligrams per deciliter [mg/dL], or corrected calcium greater than the upper limit of normal [ULN]) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Active or untreated central nervous system (CNS) metastases
* Pregnancy or breastfeeding, or intending to become pregnant during the study

Exclusion Criteria based on Organ Function or Medical History

Cardiovascular

Patients who meet the following cardiovascular exclusion criterion will be excluded from study entry:

* Left ventricular ejection fraction (LVEF) below the institutional lower limit of normal or <50%, whichever is lower

Infections Patients who meet any of the following infection exclusion criteria will be excluded from study entry:

* Positive human immunodeficiency virus (HIV) test at screening
* Active hepatitis B virus (HBV) infection (chronic or acute)
* Active hepatitis C virus (HCV) infection
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (6):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Kansas City - Menorah Medical Center, Kansas City, Kansas
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering - Basking Ridge, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- AZ Groeninge, Kortrijk, Belgium
- Germany (2):
  - Universitatsklinik Heidelberg; Universitätshautklinik und Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Universitätsklinikum Tübingen; Klinik für Urologie, Tübingen
- Hungary (3):
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Jósa András Oktatókórház, Nyíregyháza
- South Korea (4):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Yonsei Cancer Center, Seoul
- United Kingdom (3):
  - Barts & London School of Med; Medical Oncology, London
  - Royal Marsden Hospital - Fulham, London
  - The Royal Marsden, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place in six countries: Republic of Korea, Belgium, Germany, United Kingdom, Hungary and United States. No participants were enrolled in Cohort 7. Participants in long term follow up and who continued to receive treatment(s) in a post-trial access program are designated in Participant Flow as "Study terminated by Sponsor".
Pre-assignment Details: Participants with advanced solid tumors were included in the study: squamous cell carcinoma of head and neck (SCCHN), urothelial carcinoma (UC), and renal cell carcinoma (RCC).
Groups:
- Cohort 1 - SCCHN - Treatment Naive: In participants with recurrent or advanced / metastatic squamous cell carcinoma of the head and neck (SSCHN) who were anti-PD-1 and anti-PD-L1 treatment naive, cobimetinib was administered at the approved dose and schedule of 60 mg once daily (QD) for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle.
- Cohort 2 - UC - Treatment Naive: In participants with advanced / metastatic urothelial carcinoma (UC) who were anti-PD-1 and anti-PD-L1 treatment naive, cobimetinib was administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by IV infusion on Days 1 and 15 of each 28-day cycle.
- Cohort 3 - RCC - Treatment Naive: In participants with metastatic renal cell carcinoma (RCC) who were anti-PD-1 and anti-PD-L1 treatment naive, cobimetinib was administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by IV infusion on Days 1 and 15 of each 28-day cycle.
- Cohort 4 - SCCHN - Previous Treatment Exposure: In participants with SCCHN whose disease had progressed while receiving anti-PD-1 or anti-PD-L1 therapy, cobimetinib was administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by IV infusion on Days 1 and 15 of each 28-day cycle.
- Cohort 5 - UC - Previous Treatment Exposure: In participants with UC whose disease had progressed while receiving anti-PD-1 or anti-PD-L1 therapy, cobimetinib was administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by IV infusion on Days 1 and 15 of each 28-day cycle.
- Cohort 6 - RCC - Previous Treatment Exposure: In participants with RCC whose disease had progressed while receiving anti-PD-1 or anti-PD-L1 therapy, cobimetinib was administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by IV infusion on Days 1 and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
Started | 20 | 20 | 17 | 20 | 7 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 20 | 20 | 17 | 20 | 7 | 3
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 12 | 12 | 8 | 10 | 6 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 5 | 5 | 8 | 5 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure | Total
Number analyzed (Participants) | 20 | 20 | 17 | 20 | 7 | 3 | 87
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 12 | 6 | 10 | 12 | 3 | 1 | 44
  From 65-84 years | 8 | 13 | 7 | 8 | 4 | 2 | 42
  Missing | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 6 | 1 | 2 | 2 | 21
  Male | 18 | 12 | 11 | 19 | 5 | 1 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 20 | 17 | 19 | 7 | 2 | 80
  Unknown or Not Reported | 5 | 0 | 0 | 1 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 10 | 10 | 0 | 2 | 0 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 18 | 10 | 7 | 20 | 5 | 3 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate was defined as the percentage of participants with a complete response (CR) or a partial response (PR) on two consecutive tumor assessments ≥4 weeks apart, as determined by the investigators using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). CR was defined as disappearance of all lesions. PR was defined as ≥30% decrease in the sum of diameters of target lesions, in the absence of CR, new lesions, and unequivocal progression in non-target lesions.
Time Frame: Up to approximately 31 months
Population: The intent-to-treat (ITT) population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
Number analyzed (Participants) | 20 | 20 | 17 | 20 | 7 | 3
percentage of participants | 20.0 [0.00 to 40.03] | 30.0 [7.42 to 52.58] | 17.6 [0.00 to 38.71] | 0 [0.00 to 2.50] | 0 [0.00 to 7.14] | 0 [0.00 to 16.67]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from enrollment to death from any cause. The median for OS is Kaplan-Meier estimate. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Up to approximately 31 months
Population: The ITT population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
Number analyzed (Participants) | 20 | 20 | 17 | 20 | 7 | 3
months | 16.8 [6.9 to 25.8] | 18.7 [11.0 to 26.2] | 21.7 [17.4 to NA] — NA=not estimable | 7.7 [4.0 to NA] — NA=not estimable | 5.9 [3.1 to 12.5] | NA [5.9 to NA] — NA=not estimable

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from enrollment to the first occurrence of disease progression as determined by the investigator(s), using RECIST v1.1, or to death from any cause, whichever occurs first. Disease progression was defined as ≥20% increase in in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions.
Time Frame: Up to approximately 31 months
Population: The ITT population included all participants enrolled in the study.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
Number analyzed (Participants) | 20 | 20 | 17 | 20 | 7 | 3
months | 5.5 [2 to 26] | 3.4 [2 to 26] | 3.4 [1 to 28] | 3.6 [0 to 9] | 2.1 [1 to 4] | 2.7 [1 to 4]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented, confirmed objective response to disease progression as determined by the investigator, using RECIST v1.1, or to death from any cause, whichever occurs first. Objective response was defined as a complete response (CR) or a partial response (PR) on two consecutive tumor assessments ≥4 weeks apart. CR was defined as disappearance of all lesions. PR was defined as ≥30% decrease in the sum of diameters of target lesions, in the absence of CR, new lesions, and unequivocal progression in non-target lesions. Disease progression was defined as ≥20% increase in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions. Presented here is median DOR at the time of primary analysis. The median for the duration of response is Kaplan-Meier estimate. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Up to approximately 22 months
Population: ITT population: all participants enrolled in the study. Median DOR is presented at the time of primary analysis. DOR analyses were not performed at final analysis because Kaplan-Meier was not estimable at primary analysis due to too few events in Cohorts 1 and 3. There were no subsequent events in Cohorts 1 and 3. Cohorts 4-6 had no events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
Number analyzed (Participants) | 20 | 20 | 17 | 0 | 0 | 0
days | NA [NA to NA] — NA=not estimable: Kaplan-Meier was not estimable because there were too few events in Cohort 1. | 149.0 [125.0 to 173.0] | NA [NA to NA] — NA=not estimable: Kaplan-Meier was not estimable because there were too few events in Cohort 3. |  |  |

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a complete response (CR), a partial response (PR), or stable disease at 16 weeks as determined by the investigator using RECIST v1.1. CR was defined as disappearance of all lesions. PR was defined as ≥30% decrease in the sum of diameters of target lesions, in the absence of CR, new lesions, and unequivocal progression in non-target lesions. Stable disease was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for disease progression. Disease progression was defined as ≥20% increase in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions.
Time Frame: At 16 weeks
Population: The ITT population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
Number analyzed (Participants) | 20 | 20 | 17 | 20 | 7 | 3
percentage of participants | 50.0 [25.59 to 74.41] | 40.0 [16.03 to 63.97] | 23.5 [0.42 to 46.63] | 25.0 [3.52 to 46.48] | 0 [0.00 to 7.14] | 0 [0.00 to 16.67]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to approximately 31 months
Population: The safety population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
Number analyzed (Participants) | 20 | 19 | 17 | 20 | 7 | 3
participants | 20 | 19 | 17 | 20 | 7 | 3

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Cobimetinib
Description: Cmax is the maximum (or peak) concentration that a study drug achieves in the body.
Time Frame: Day 15 of Cycle 3 (cycle is 28 days): 2-4 hours after cobimetinib dose
Population: Pharmacokinetic (PK) analysis population consisted of participants with sufficient data to enable estimation of key parameters, with participants grouped according to treatment received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Cohorts 1-6: In all participants cobimetinib was administered at the approved dose and schedule of 60 mg QD for 21 days and 7 days off of each 28-day cycle; and atezolizumab 840 mg by IV infusion on Days 1 and 15 of each 28-day cycle.
Arm/Group | Cohorts 1-6
Number analyzed (Participants) | 33
nanogram per milliliter (ng/mL) | 285 (56.5)

8. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Cobimetinib
Description: Cmin is the minimum (or trough) concentration that a study drug achieves in the body.
Time Frame: Day 15 of Cycle 3 (cycle is 28 days): prior to cobimetinib dose
Population: PK analysis population consisted of participants with sufficient data to enable estimation of key parameters, with participants grouped according to treatment received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohorts 1-6
Number analyzed (Participants) | 30
ng/mL | 174 (152)

9. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab
Description: Cmax is the maximum (or peak) concentration that a study drug achieves in the body.
Time Frame: 30 minutes following end of atezolizumab infusion on Day 15 of Cycle 3 (each cycle is 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohorts 1-6
Number analyzed (Participants) | 40
ng/mL | 417000 (50.2)

10. Secondary Outcome: Minimum Serum Concentration (Cmin) of Atezolizumab
Description: Cmin is the minimum (or trough) concentration that a study drug achieves in the body.
Time Frame: Prior to atezolizumab infusion on Day 1 of Cycles (each cycle is 28 days) 2, 4, 8, 12, and 16, Day 15 of Cycle 3
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohorts 1-6
Number analyzed (Participants) | 61
ng/mL | 112000 (219)

11. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs)
Description: Participants were considered to be ADA positive if they were missing data at baseline but developed an ADA response following study drug administration (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post-baseline samples was at least 4-fold greater (i.e., ≥0.60-titer units) than the titer of the baseline sample (treatment-enhanced ADA response). Participants were considered to be ADA negative if they were missing data at baseline, had a post-baseline ADA result, and all post-baseline samples were negative, or if they were ADA positive at baseline but did not have any post-baseline samples with a titer that was at least 4-fold greater than the titer of the baseline sample (treatment unaffected).
Time Frame: Day 1 of Cycles (each cycle is 28 days) 1, 2, 4, 8, 12, and 16; Day 15 of Cycle 3; at atezolizumab treatment discontinuation visit, and <90 days after last atezolizumab infusion (up to approximately 31 months)
Population: The safety population included all enrolled participants who received at least one dose of study drug. Number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
Number analyzed (Participants) | 19 | 19 | 17 | 10 | 1 | 2
Participants | 1 | 10 | 6 | 5 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to approximately 31 months
Description: The safety population included all enrolled participants who received at least one dose of study drug.
Arm/Group | Cohort 1 - SCCHN - Treatment Naive | Cohort 2 - UC - Treatment Naive | Cohort 3 - RCC - Treatment Naive | Cohort 4 - SCCHN - Previous Treatment Exposure | Cohort 5 - UC - Previous Treatment Exposure | Cohort 6 - RCC - Previous Treatment Exposure
All-Cause Mortality (participants affected / at risk) | 12/20 | 12/19 | 8/17 | 12/20 | 6/7 | 1/3
Serious Adverse Events (participants affected / at risk) | 13/20 | 9/19 | 8/17 | 10/20 | 4/7 | 1/3
Other Adverse Events (participants affected / at risk) | 20/20 | 19/19 | 17/17 | 19/20 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - SCCHN - Treatment Naive (N=20) | Cohort 2 - UC - Treatment Naive (N=19) | Cohort 3 - RCC - Treatment Naive (N=17) | Cohort 4 - SCCHN - Previous Treatment Exposure (N=20) | Cohort 5 - UC - Previous Treatment Exposure (N=7) | Cohort 6 - RCC - Previous Treatment Exposure (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
IMMUNE-MEDIATED HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE RESPIRATORY FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IMMUNE-MEDIATED ENCEPHALITIS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEPHRITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROSTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - SCCHN - Treatment Naive (N=20) | Cohort 2 - UC - Treatment Naive (N=19) | Cohort 3 - RCC - Treatment Naive (N=17) | Cohort 4 - SCCHN - Previous Treatment Exposure (N=20) | Cohort 5 - UC - Previous Treatment Exposure (N=7) | Cohort 6 - RCC - Previous Treatment Exposure (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 8 (9) | 6 (6) | 4 (5) | 2 (4) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INNER EAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
THYROIDITIS (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHORIORETINOPATHY (Eye disorders) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
ENTROPION (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYELID OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MACULAR OEDEMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPTIC NERVE DISORDER (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIORBITAL OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RETINAL OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETINOPATHY (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBRETINAL FLUID (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SWELLING OF EYELID (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRICHIASIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VITREOUS FLOATERS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2) | 1 (3) | 2 (3) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANGULAR CHEILITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 5 (7) | 3 (3) | 4 (4) | 1 (2) | 0 (0)
DIAPHRAGMATIC HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 7 (9) | 11 (15) | 9 (13) | 13 (16) | 5 (6) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GLOSSITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GLOSSODYNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIP OEDEMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
LIP PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIP SWELLING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MUCOUS STOOLS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 3 (3) | 5 (5) | 6 (8) | 4 (5) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL DISCHARGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 2 (3) | 5 (5) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 7 (9) | 4 (8) | 3 (3) | 4 (4) | 1 (2) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
FACE OEDEMA (General disorders) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
FACIAL PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 6 (6) | 9 (14) | 5 (7) | 5 (5) | 5 (5) | 0 (0)
GENERALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOCALISED OEDEMA (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
OEDEMA (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
PAIN (General disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 7 (9) | 5 (9) | 1 (1) | 4 (4) | 0 (0)
SWELLING FACE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONGUE FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STRESS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 3 (3) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 4 (4) | 7 (9) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD MAGNESIUM DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD URIC ACID INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLATELET COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN B12 DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN D DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 2 (3) | 3 (3) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (4) | 7 (8) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRISMUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CAUDA EQUINA SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS POSTURAL (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TASTE DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANGER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCROTAL OEDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TESTICULAR SWELLING (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RALES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 2 (3) | 0 (0)
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (5) | 1 (2) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERTRIGO (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (2) | 4 (4) | 3 (6) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 9 (10) | 9 (11) | 12 (14) | 5 (6) | 5 (7) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (8) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT03264066/Prot_SAP_000.pdf